CLINICAL TRIAL: NCT05806788
Title: Binge Eating Syndrome Treatment for Older Women (BESTOW)
Acronym: BESTOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Lisa Kilpela, Associate Professor, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC20220898H; 5K76AG060003 (NIH)
Record Dates: First submitted 2023-03-22; First posted 2023-04-10 (Actual); Results first posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Binge Eating
Keywords: Binge Eating Spectrum; Cognitive-behavioral therapy; Body Image
MeSH Terms: conditions — Bulimia

STUDY DESIGN:
Intervention Model Description: This study is a beta-testing of a new behavioral intervention treatment - all participants will be assigned to the treatment and give feedback on the treatment throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BESTOW behavioral intervention (Experimental): The intervention will utilize behavioral-based strategies to reduce BE and improve health behaviors, with content including strategies to improve body image, regulation of eating behaviors, and integration of physical activity with an emphasis on body function, health, and longevity.
  Interventions: Behavioral: Binge Eating Syndrome Treatment (BESTOW)

INTERVENTIONS:
Behavioral: Binge Eating Syndrome Treatment (BESTOW) — The BESTOW program involves discussions as well as written and behavioral activities. Participants will also be asked to complete activities, or 'homework,' in between sessions that will help to stop binge eating and to improve eating habits.

SUMMARY:
Twenty women, ages 60 or older, will be consented and enrolled in a single-arm, pilot implementation trial of the age-tailored cognitive-behavioral based BE intervention. Participants will complete assessments at baseline, post-intervention, and at two follow-up timepoints; weekly BE frequency will be collected to monitor progress during the intervention period.

DETAILED DESCRIPTION:
The intervention being studied will be an age-tailored, cognitive-behavioral therapy (CBT) based behavioral intervention for binge eating (BE), delivered by the PI, a licensed clinical psychologist, in small group format (4-6 participants per group) over 12-16 weeks. The intervention will utilize behavioral-based strategies to reduce BE and improve health behaviors, with content including strategies to improve body image, regulation of eating behaviors, and integration of physical activity with an emphasis on body function, health, and longevity. The final session number, frequency, content, and timeline will be determined during intervention-tailoring process not a part of this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age 60 years and over
* Binge eating (BE) ≥1/week during the past ≥3 months
* Community-dwelling
* Able to provide informed consent
* Consistent medication regimen for 3 months

Exclusion Criteria:

* Significant cognitive impairment
* Nursing home, long-term care facility
* Psychosis or imminent suicide risk
* Current BE treatment

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Kilpela, PhD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Per guidelines, we will publish deidentified data results from this trial via ClinicalTrials.gov within one year of study completion. Participants will be informed of this at the time of consent, if they are interested in learning the results from the study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within one year of study completion

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BESTOW Behavioral Intervention
Started | 20
Completed | 17
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | BESTOW Behavioral Intervention
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (4.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Feasibility - Usage Rating Profile - Intervention
Description: Score on the Feasibility Usage Rating Profile. This scale gathers patient reported feasibility of the intervention (e.g., time needed, quality of materials, simplicity of the intervention) to be completed after doing the intervention. This scale has six items; total scores range from 1-6 and a higher scores indicate greater feasibility.
Time Frame: 6 weeks (post), and 2 month follow-up
Population: Post-assessment completers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BESTOW Behavioral Intervention
Number analyzed (Participants) | 17
score on a scale
  6 weeks (Post intervention) | 5.44 (0.85)
  2-month follow-up | 5.53 (0.83)

2. Primary Outcome: Acceptability - Usage Rating Profile - Intervention
Description: Score on the Acceptability Usage Rating Profile scale which gathers participant ratings of how acceptable the treatment is for targeting binge eating (e.g., how helpful the intervention was, how much they liked it, willingness to do the intervention) to be completed after doing the intervention. This scale has eight items; total scores range from 1-6, a higher score indicates greater acceptability.
Time Frame: 6 weeks (post), and 2 month follow-up
Population: Post-assessment completers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BESTOW Behavioral Intervention
Number analyzed (Participants) | 17
score on a scale
  6 weeks (post assessment) | 5.58 (0.75)
  2-month follow-up | 5.50 (0.76)

3. Secondary Outcome: Binge Eating Score (BES)
Description: Change in score on the BES survey. The BES is a 16-item, self-report survey that assess binge eating. Total scores range from 0 to 46, with higher scores meaning more severe binge eating symptoms (Gormally et al., 1982).
Time Frame: Baseline, 6 weeks, 1 month, and 2 month follow-up
Population: Completers. One of the subjects was too busy to complete the questionnaire at the 1 month follow up, so only 16 participants were evaluable at that time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BESTOW Behavioral Intervention
Number analyzed (Participants) | 20
score on a scale
  Baseline | 24.78 (5.89)
  Post: number analyzed (Participants) | 17
  Post | 14.81 (5.87)
  1-month follow-up: number analyzed (Participants) | 16
  1-month follow-up | 13.24 (6.64)
  2-month follow-up: number analyzed (Participants) | 17
  2-month follow-up | 13.81 (9.08)

4. Secondary Outcome: Geriatric Depression Scale Score (Center for Epidemiologic Studies-Depression Scale; CES-D)
Description: The CES-D is a 10-item, self-report survey that assess depressive symptoms. Mean scores range from 0 to 3, with higher scores indicating more depressive symptoms (Lewinsohn et al., 1997).
Time Frame: Baseline, 6 weeks (post), 1 month, and 2 month follow-up
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BESTOW Behavioral Intervention
Number analyzed (Participants) | 20
score on a scale
  Baseline | 1.15 (0.59)
  Post: number analyzed (Participants) | 17
  Post | 0.91 (0.75)
  1-month follow-up: number analyzed (Participants) | 16
  1-month follow-up | 0.93 (0.69)
  2-month follow-up: number analyzed (Participants) | 17
  2-month follow-up | 1.00 (0.81)

ADVERSE EVENTS:
Time Frame: Baseline to 2-month follow-up
Description: Definitions did not differ from clinicaltrials.gov
Arm/Group | BESTOW Behavioral Intervention
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-10): https://cdn.clinicaltrials.gov/large-docs/88/NCT05806788/Prot_SAP_001.pdf
  • Informed Consent Form (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT05806788/ICF_000.pdf